CLINICAL TRIAL: NCT02095262
Title: Auditory Games for Tinnitus Benefit: Interactive Versus Reactive Auditory Discrimination Games
Brief Title: Gameplay as a Source of Intrinsic Motivation in a Randomized Controlled Trial of Auditory Training for Tinnitus
Acronym: TAG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11IH001
Record Dates: First submitted 2014-03-08; First posted 2014-03-24 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- STAR2 (Active Comparator): Reactive auditory training
  Interventions: Other: reactive auditory training
- Treasure Hunter (Experimental): Interactive auditory training
  Interventions: Other: Interactive auditory training
- Submarine (Experimental): Interactive auditory training
  Interventions: Other: Interactive auditory training

INTERVENTIONS:
Other: reactive auditory training
  Arms: STAR2
Other: Interactive auditory training
  Arms: Submarine; Treasure Hunter

SUMMARY:
Tinnitus refers to a the perception of a ringing, hissing or buzzing sound despite there being no such sound in the external world. It is prevalent and for many individual is a distressing condition. Recent advances in the understanding of changes in the hearing brain and their relation to tinnitus perception has led to a focus on forms of active auditory training which might provide effective techniques for tinnitus management. Our recent trial of auditory training provided evidence that training using sounds where there is no hearing loss has benefit in terms of reduced tinnitus intrusiveness, above training at where there is some level of hearing loss. Our next challenge is to build on this finding in ways that might maximize the benefits we observe.

The training software we used previously was developed for use with children. Past participants have given mixed reviews of this software. While some enjoyed the training or found it soporific, others reported that they found it too monotonous and un-motivating. We therefore wish to explore the impact of different game mechanics in the delivery of auditory training and have designed two different interactive games in the context of training for tinnitus benefit. These games will deliver the same type of auditory training as the software we currently use, but should be intrinsically motivating, i.e. be a game that the people are motivated to play irrespective of any potential benefit for tinnitus. The game we previously used is reactive, i.e. the sounds play and the player selects what they think is the correct answer (odd one out).

The two new games we wish to test can be described as interactive, i.e. players control the sound delivery and actively seek the correct answer: this may have additional benefit for tinnitus.

ELIGIBILITY:
Inclusion Criteria:

(i) Chronic subjective tinnitus (experienced for over 6 months)

(ii) Aged 18 + years old

(iii) Not currently receiving treatment for tinnitus from the National Health Service or other sources

Exclusion Criteria:

(i) Significant distress (Beck anxiety score >25, Beck depression score >13)

(ii) Hyperacusis (Khalfa Hyperacusis Questionnaire score >27)

(iii) Significant bilateral hearing loss (>39 decibel at all tested frequencies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Questionnaire | 4 weeks
  Two pre-intervention assessments & post intervention

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory | 6 weeks
  Two pre-intervention assessments & post intervention
psychoacoustic measures of tinnitus | 4 weeks
  Pre and post intervention measure

OTHER OUTCOMES:
Test of Everyday Attention | 4 weeks
  Pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Hall, Professor, Principal Investigator — University of Nottingham
Locations (1):
- NIHR Nottingham Hearing Biomedical Research Unit, Nottingham, United Kingdom

REFERENCES:
- [Result] Hoare DJ, Van Labeke N, McCormack A, Sereda M, Smith S, Al Taher H, Kowalkowski VL, Sharples M, Hall DA. Gameplay as a source of intrinsic motivation in a randomized controlled trial of auditory training for tinnitus. PLoS One. 2014 Sep 12;9(9):e107430. doi: 10.1371/journal.pone.0107430. eCollection 2014. PMID 25215617
- [Derived] Sereda M, Edmondson-Jones M, Hall DA. Relationship between tinnitus pitch and edge of hearing loss in individuals with a narrow tinnitus bandwidth. Int J Audiol. 2015 Apr;54(4):249-56. doi: 10.3109/14992027.2014.979373. Epub 2014 Dec 3. PMID 25470623